CLINICAL TRIAL: NCT03450720
Title: Evaluation of the Pharmacokinetics, Safety and Tolerability of a Single Dose of GLPG2737 Administered as Oral Suspension in Male Subjects With Cystic Fibrosis
Brief Title: Pharmacokinetics of GLPG2737 in Male Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLPG2737-CL-104; 2017-000449-38 (EudraCT Number)
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLPG2737 single dose. (Experimental): Single dose of GLPG2737 oral suspension.
  Interventions: Drug: GLPG2737 single dose

INTERVENTIONS:
Drug: GLPG2737 single dose — GLPG2737 oral suspension, single dose

SUMMARY:
This is a single dose, open label study in adult male subjects with cystic fibrosis to investigate the pharmacokinetics, safety and tolerability of GLPG2737.

ELIGIBILITY:
Inclusion Criteria:

* Male subject ≥18 years of age on the day of signing the informed consent form (ICF).
* A confirmed clinical diagnosis of CF.
* Two mutations in the cystic fibrosis transmembrane conductance regulator (CFTR) gene belonging to class I and/or class II and/or class III (documented in the subject's medical record or CF registry).
* Weight ≥40 kg.
* Exocrine pancreatic insufficiency (documented in the subject's medical record).
* Stable concomitant medication regimen for at least 2 weeks prior to study drug administration.
* Forced expiratory volume in one second (FEV1) ≥40% of predicted normal for age, gender and height at screening (pre- or postbronchodilator).

Exclusion Criteria:

* History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
* Unstable pulmonary status or respiratory tract infection (including rhinosinusitis) requiring a change in therapy within 2 weeks prior to study drug administration.
* History of hepatic cirrhosis with portal hypertension (e.g.,signs/symptoms of splenomegaly, esophageal varices).
* Use of CFTR modulator therapy (e.g., lumacaftor or ivacaftor) within 2 weeks prior to study drug administration.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG2737and its metabolite. | Between day 1 pre-dose and 48 hours post-dose.
  To characterize the PK of GLPG2737 and its metabolite after a single oral dose in CF subjects.
Time of occurrence of Cmax for GLPG2737(tmax) | Between day 1 pre-dose and 48 hours post-dose.
  To determine PK parameters of GLPG2737 and its metabolite after given a single oral dose in CF subjects.
Plasma concentration observed at 24 hours post-dos (C24h) | Between day 1 pre-dose and 48 hours post-dose.
  To assess PK parameters of GLPG2737 and its metabolite after given a single oral dose in CF subjects.
Area under the plasma concentration-time curve for GLPG2737 (AUC0-24h) | Between day 1 pre-dose and 48 hours post-dose.
  To determine the PK of GLPG2737 and its metabolite after a single oral dose in CF subjects.
Area under the plasma concentration-time curve from time zero until 48 hours post-dose (AUC0-48h) | Between day 1 pre-dose and 48 hours post-dose.
  To determine the PK of GLPG2737 and its metabolite after a single oral dose in CF subjects.
Terminal plasma elimination rate constant (ke) | Between day 1 pre-dose and 48 hours post-dose.
  To determine the PK of GLPG2737 and its metabolite after a single oral dose in CF subjects.
Apparent terminal elimination half-life ( t1/2) | Between day 1 pre-dose and 48 hours post-dose.
  To determine the PK of GLPG2737 and its metabolite after a single oral dose in CF subjects.

SECONDARY OUTCOMES:
Number of subjects with adverse events. | Between screening and 15 days post-dose
  To determine the safety and tolerability of GLPG2737 after a single oral dose in CF subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van de Steen, MD MBA, Study Director — Galapagos NV
Locations (1):
- UZ KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided